CLINICAL TRIAL: NCT01636258
Title: Diet, Exercise, Cooking, and Stress Management for Patients With Prediabetes: A Pilot Randomized Controlled Study
Brief Title: FRESH Study (Fitness, Relaxation and Eating to Stay Healthy)
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-340
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Prediabetes; Overweight
Keywords: Prediabetes; Overweight; African American; Women; Cooking; Nutrition; Exercise; Stress Management
MeSH Terms: conditions — Prediabetic State; Overweight; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Control group (No Intervention): These participants will continue to receive their usual care from their primary medical care team.
- Arm B (Experimental): Arm includes diet instruction, exercise, stress management, and culinary education
  Interventions: Behavioral: Stress Management; Behavioral: Diet; Behavioral: Exercise; Behavioral: Culinary education

INTERVENTIONS:
Behavioral: Stress Management — Every other week
  Arms: Arm B
Behavioral: Diet — Every other week
  Arms: Arm B
Behavioral: Exercise — Every week
  Arms: Arm B
Behavioral: Culinary education — Every other week
  Arms: Arm B

SUMMARY:
To examine whether a lifestyle program results in weight loss and thereby delays or prevents progression of pre-diabetes to diabetes, we propose a pilot randomized controlled trial of 6 weeks duration with 30 participants held at Stephanie Tubbs Jones Health Center. Participants are randomized to receive all of the following: nutrition education, exercise instruction, stress management instruction, and culinary education or follow usual care. Outcomes include: blood sugars and cholesterol, weight, waist circumference, blood pressure, diet, physical activity, perceived stress, and class attendance. Analysis is by Intention to treat analysis of variance. Results will be used to help design larger randomized trial in the future.

DETAILED DESCRIPTION:
Control group:

These participants will continue to receive their usual care from their primary medical care team.

Intervention group:

The participants will receive nutrition education, exercise instruction, stress management instruction,and culinary education

ELIGIBILITY:
Inclusion Criteria:

* Study participants must:

  1. Be capable of giving informed consent
  2. Understand and voluntarily sign the informed consent form.
  3. Be females at least 18 years of age and identify themselves as African-American
  4. Have prediabetes as defined by the American Diabetes Association: history of glycated hemoglobin (HgbA1c) 5.7-6.4 % or fasting blood glucose 100-125 mg/dL (5.6-6.9 mmol/L) (fasting defined as no caloric intake for at least 8 hours), or a 2-hour plasma glucose 140-199 mg/dL (7.8-11.0 mmol/L) during an oral glucose tolerance test (as described by the World Health Organization using a glucose load of 75 g anhydrous glucose dissolved in water)
  5. Have a body mass index (BMI, defined as weight in kilograms divided by height in meters squared) greater than or equal to 25

Exclusion Criteria:

1. Current or previous diagnosis of diabetes or a history of HgbA1c ≥ 6.5% or fasting blood glucose ≥ 126 mg/dL (7.0 mmol/L) (fasting defined as no caloric intake for at least 8 hours), or a 2-hour plasma glucose ≥ 200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test or a history of classic symptoms of hyperglycemia or hyperglycemic crisis and a random plasma glucose ≥ 200 mg/dL (11.1 mmol/L).
2. Normal glycemia or a currently with a HgbA1c < 5.7% or fasting blood glucose < 100 mg/dL (7.0 mmol/L) (fasting defined as no caloric intake for at least 8 hours), or a 2-hour plasma glucose < 140 mg/dL (11.1 mmol/L) during an oral glucose tolerance test
3. Current or past use of oral hypoglycemic agents (including, but not limited to, metformin, rosiglitazone, pioglitazone, glipizide, and glyburide) or insulin
4. Male gender
5. History of congestive heart failure
6. History of renal failure, dialysis, or creatinine greater than 2 mg/dL
7. History of liver failure or a liver dysfunction with a increase by a factor of 2 above the upper limit of normal in alanine aminotransferase or aspartate aminotransferase
8. History of gastrointestinal disorder that would prevent adherence to the recommended diet (e.g. celiac disease, inflammatory bowel disease, history of bariatric surgery, history of intestinal surgery)
9. Presence of active cancer
10. History of coronary artery disease or cerebrovascular disease
11. History of uncontrolled hypertension
12. Participation in another lifestyle modification trial
13. Pregnancy or lactating or planning to be pregnant
14. Current alcoholism or abuse of recreational drugs
15. Hospitalization for depression in past 12 months
16. Travel plans that do not permit full participation or participant lives too far from Health Center to permit full participation
17. History of bariatric surgery, small bowel resection, or extensive bowel resection
18. Chronic treatment with systemic steroids
19. Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
20. Inability to walk two blocks
21. Other medial, psychiatric, or behavioral limitations that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention protocol
22. Amputation of lower limb for nontraumatic causes
23. Self report of HIV-positivity or active tuberculosis
24. Documented history of pulmonary embolus in past six months
25. Chronic obstructive pulmonary disease that would limit ability to follow the study protocol
26. Self-reported chronic hepatitis B or C or cirrhosis; inflammatory bowel disease requiring treatment in past year; Cushing's syndrome; acromegaly (clinical diagnosis or self-report); any major organ transplant
27. Unwilling or uninterested in participating in group lifestyle education sessions
28. Current regular corticosteroid use
29. Active polycystic ovarian syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Bernstein, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Stephanie Tubbs Jones Health Center, East Cleveland, Ohio, United States

REFERENCES:
- [Derived] Bernstein AM, Gendy G, Rudd N, Doyle J, Fay S, Moffett K, Morrison S, Bena J, Cotey S, Roizen MF, Golubic M. Management of prediabetes through lifestyle modification in overweight and obese African-American women: the Fitness, Relaxation, and Eating to Stay Healthy (FRESH) randomized controlled trial. Public Health. 2014 Jul;128(7):674-7. doi: 10.1016/j.puhe.2014.04.005. Epub 2014 Jul 2. No abstract available. PMID 24996961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May and August, 2012. Recruitment methods included flyers distributed to health centers, libraries, and community health outreach events; advertisements in Cleveland Clinic and Community newsletters; and a television appearance on popular Sunday morning news program by one of the research team members.
Pre-assignment Details: Two participants who were enrolled in study were excluded at baseline laboratory check due to glycated hemoglobin (HgbA1c) value below 5.7%.
Groups:
- Arm B: Intervention Group: Arm includes diet instruction, exercise, stress management, and culinary education
  Exercise : Every week
  Diet : Every other week
  Culinary education : Every other week
  Stress Management : Every other week
Period: Overall Study
Arm/Group | Arm A: Control Group | Arm B: Intervention Group
Started | 13 | 14
Completed | 12 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Control Group | Arm B: Intervention Group | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (9.3) | 57.7 (11.4) | 55 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Effect of "FRESH" Program on Weight Loss
Description: Change in weight measured at baseline and followup (at 8-14 weeks).
Time Frame: Baseline line and final followup visit (at 8-14 weeks)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm A: Control Group | Arm B: Intervention Group
Number analyzed (Participants) | 12 | 14
kg | -0.5 (2.0) | -0.2 (2.2)
Statistical Analysis 1: Comparison: Arm A: Control Group vs Arm B: Intervention Group; No sample size calculation performed since it was a pilot study. Null hypothesis was no difference between groups; Test type: Superiority or Other; p = 0.72, t-test, 2 sided — P-value less than 0.05 considered statistically significant a priori. No multiple comparison adjustment made; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.4 to 2.0], Standard Deviation 2.1

2. Secondary Outcome: Diet - Daily Calorie Intake
Description: Change in daily caloric intake as measured by online 24-hour recall dietary program
Time Frame: Baseline and final followup visit (at 8-14 weeks)
Measure: Mean (Inter-Quartile Range); unit: Kcal/day
Arm/Group | Arm A: Control Group | Arm B: Intervention Group
Number analyzed (Participants) | 12 | 14
Kcal/day | 172.2 [-347.4 to 939] | 36.5 [-266.7 to 459]
Statistical Analysis 1: Comparison: Arm A: Control Group vs Arm B: Intervention Group; No sample study calculation performed since it was a pilot study. Null hypothesis was no difference between groups; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Exercise
Description: Change in 7-day average steps/day as measured by pedometer at baseline and followup (at 8-14 weeks).
Time Frame: Baseline and final followup visits (at 8-14 weeks)
Measure: Mean (Inter-Quartile Range); unit: steps/day
Arm/Group | Arm A: Control Group | Arm B
Number analyzed (Participants) | 12 | 14
steps/day | -1290 [-2932.3 to 503] | 253.4 [-903.9 to 1201]
Statistical Analysis 1: Comparison: Arm A: Control Group vs Arm B; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Stress
Description: Change of Psychosocial Stress (PSS-10) scores (total range 0-40) measured at baseline and followup (at 8-14 weeks). Higher score reflects worse outcome.
Time Frame: baseline and followup visit (at 8-14 weeks)
Measure: Mean (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Arm A: Control Group | Arm B
Number analyzed (Participants) | 12 | 14
scores on a scale | 0.5 [-2.0 to 2.0] | -1.0 [-3.0 to 4.0]
Statistical Analysis 1: Comparison: Arm A: Control Group vs Arm B; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Sleep
Description: Change in self-reported average hours of sleep/night measured at baseline and followup (at 8-14 weeks).
Time Frame: baseline and followup visit (at 8-14 weeks)
Measure: Mean (Inter-Quartile Range); unit: hours/night
Arm/Group | Arm A: Control Group | Arm B
Number analyzed (Participants) | 12 | 14
hours/night | 0.0 [0.0 to 1.0] | 0.0 [-1.0 to 0.0]

ADVERSE EVENTS:
Time Frame: 6 week intervention program
Description: Serious and other (non-serious) adverse events were collected/assessed, but none observed.
Arm/Group | Arm A: Control Group | Arm B: Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No